CLINICAL TRIAL: NCT04449614
Title: A Review of Surgical Management of Congenital Pulmonary Airway Malformations (CPAM): A Decade of Experience
Acronym: CPAM
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 238420
Record Dates: First submitted 2018-10-10; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Arteriovenous Malformation; Congenital Disorders
MeSH Terms: conditions — Pulmonary Arteriovenous Fistulas; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Inclusion criteria: All consenting Infants and children who have had A Congenital Pulmonary Airway Malformation (CPAM) surgically removed by thoracoscopy over a 10 year period (2008-2017) in a regional centre.
  Exclusion criteria: Non consenting participants
  Interventions: Procedure: Thoracoscopic CPAM resection

INTERVENTIONS:
Procedure: Thoracoscopic CPAM resection — Surgical removal of lung lesion

SUMMARY:
Congenital pulmonary malformation in children is a rare abnormality mostly diagnosed before birth during antenatal ultrasound examinations. These lesions may expand to form lung cysts in children, cause recurrent lung infections and has a potential for malignant change. Therefore, surgical removal in childhood is favoured as the treatment of choice.

The surgical correction may involve 'open' surgery or 'key hole' surgery. There is, however, a variation in surgical and anaesthetic techniques and timing of this surgery and subsequent complications reported post-surgery.

The purpose of this investigation is to review anaesthetic and surgical case notes and the subsequent well-being of all children who underwent lung surgery to remove above lung lesions over the last 10 years (2008-2017) at a regional centre. The aim is to look at the current status of these children in relation to their health, growth and development evaluated via a 20-minute structured telephone interview with prior consent.

DETAILED DESCRIPTION:
Congenital pulmonary airway malformation (CPAM) (previously named congenital cystic adenomatoid malformation) is a rare abnormality, first described in 1949. CPAM results from adenomatoid proliferation of the terminal bronchioles causing cyst formation, which may impair normal alveolar growth. It occurs more commonly in males and has an estimated incidence of 1:11000 to 1:35000. Most are diagnosed on routine antenatal ultrasonography. Most involve lower lobes, occasionally lesions are bilateral. CPAM lesions are usually managed by surgical removal in childhood due to the risk of serious infection, and potential for malignant change. A recent meta-analysis has favoured surgical management.

Historically, correction of CPAM was by open thoracotomy and surgical resection. This has evolved, however, and since 2008 more than 50 surgical corrections have been carried out thoracoscopically at King's College Hospital. The perioperative anaesthetic management of these children has also evolved, with the increasing use of selective lung ventilation.

The age range at surgery is variable, usually 1 - 14 years, and just over half being asymptomatic. Anaesthetic techniques are variable: for example, the deployment of selective lung ventilation techniques, the choice of anaesthetic agents and the types of invasive monitoring. Surgical duration is typically 3-4 hours. A degree of hypercarbia occurs in most cases during the procedure because of reduced minute ventilation to facilitate surgical access, and the absorption of carbon dioxide insufflated into the pleural space. Around 1/3rd receive blood transfusions. Perioperative complications include: respiratory problems causing hypoxia, requirement for re-intubation, conversion to open thoracotomy, bradycardia, surgical emphysema and sometimes the requirement for prolonged post-operative respiratory support including ventilation, CPAP and chest drain management, bronchopulmonary fistulae, and chylothorax and rarely seizures and cerebral infarction.

In general, post-operative care includes at least 24 hours critical care and another 6-7 days in hospital. The mainstay of early post-operative pain control is either with morphine using a nurse controlled intravenous analgesia system, or with epidural analgesia. These are supplemented with oral analgesic regimens. Children who were preoperatively symptomatic seem more likely to develop perioperative complications.

Objective The purpose of this investigation is to review all children who underwent CPAM surgery over the last 10 years at a single regional centre and carry out a descriptive evaluation of pre-operative factors, anaesthetic and surgical factors, peri- and post-operative morbidity, mortality and subsequent long term outcome.

Methods A retrospective review of all CPAM resections performed since 2008 at a single centre. The data will be retrieved from electronic and paper based medical records, anaesthetics records and operation notes. A prospective analysis of the post-operative course and events will be undertaken. A detailed evaluation of these children in relation to their health, growth and development will be carried out via a structured 20-minute telephone interview with prior consent.

Analysis Outcomes will be compared across preoperatively symptomatic and asymptomatic groups using Mann-Whitney/Wilcoxon test or Student t test for continuous data or the chi square for categorical data. All tests were 2-tailed, and P< 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

All children undergoing surgery for a CPAM removal between 2008 - 2017 at a regional hospital.

Exclusion Criteria:

Lack of informed consent. Inability to contact parents/guardian for the required post-operative interview

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants and children who had undergone thoracoscopic surgery for a CPAM from 2008 to 2017 at a regional centre
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Perioperative morbidity associated with the CPAM removal surgical episode | 28 days postoperative
  This will be a descriptive measure of perioperative complications, namely, number including converted to 'open' surgery from thoracoscopy and its reasons, postoperative respiratory complications needing active therapy such as return to theatre, reintubation, insertion of chest drains to manage pneumothorax, haemothorax or chylothorax, duration of intensive care needed and duration of hospital stay needed.
Perioperative mortality associated the CPAM removal surgical episode | 28 days postoperative
  This will include 28 day mortality associated with the surgical episode

SECONDARY OUTCOMES:
Post surgery long-term well being as reported by parents/guardian | A prospective 1 year to complete a telephone follow-up of all participant children who had their surgery performed between 2007-2017
  This will be a qualitative assessment of the child's postoperative well-being as reported by the parents/guardian during hospital follow up clinics or an assessment by telephone using a standard questionnaire to assess well-being, growth and development of the child as reported by the parents or guardian. This will in addition include the frequency of any respiratory symptoms, therapeutic needs and hospitalisations encountered by the child following the removal of CPAM.
Post surgery long-term development and growth of children as reported by parent/guardian | A prospective 1 year to complete a telephone follow-up of all participant children who had their surgery performed between 2007-2017
  This will be parental opinion of child's well-being when compared to that of preoperative cognitive function, development, and general health. In summary this is a qualitative assessment of child's health as reported by the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Chulananda Goonasekera, Principal Investigator — Consultant Anaesthetist
Locations (1):
- Kings College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Subramanyam R, Ledbetter K, Fleck R, Mahmoud M. Images in Anesthesiology: Congenital Pulmonary Airway Malformation. Anesthesiology. 2017 Aug;127(2):382. doi: 10.1097/ALN.0000000000001602. No abstract available. PMID 28719530
- [Background] Cloutier MM, Schaeffer DA, Hight D. Congenital cystic adenomatoid malformation. Chest. 1993 Mar;103(3):761-4. doi: 10.1378/chest.103.3.761. PMID 8449065
- [Background] Sfakianaki AK, Copel JA. Congenital cystic lesions of the lung: congenital cystic adenomatoid malformation and bronchopulmonary sequestration. Rev Obstet Gynecol. 2012;5(2):85-93. PMID 22866187
- [Background] Mann S, Wilson RD, Bebbington MW, Adzick NS, Johnson MP. Antenatal diagnosis and management of congenital cystic adenomatoid malformation. Semin Fetal Neonatal Med. 2007 Dec;12(6):477-81. doi: 10.1016/j.siny.2007.06.009. Epub 2007 Oct 22. PMID 17950681
- [Background] David M, Lamas-Pinheiro R, Henriques-Coelho T. Prenatal and Postnatal Management of Congenital Pulmonary Airway Malformation. Neonatology. 2016;110(2):101-15. doi: 10.1159/000440894. Epub 2016 Apr 13. PMID 27070354
- [Result] Sueyoshi R, Koga H, Suzuki K, Miyano G, Okawada M, Doi T, Lane GJ, Yamataka A. Surgical intervention for congenital pulmonary airway malformation (CPAM) patients with preoperative pneumonia and abscess formation: "open versus thoracoscopic lobectomy". Pediatr Surg Int. 2016 Apr;32(4):347-51. doi: 10.1007/s00383-015-3848-z. Epub 2015 Dec 12. PMID 26661941
- [Result] CH'IN KY, TANG MY. Congenital adenomatoid malformation of one lobe of a lung with general anasarca. Arch Pathol (Chic). 1949 Sep;48(3):221-9. No abstract available. PMID 18137795
- [Result] Laberge JM, Flageole H, Pugash D, Khalife S, Blair G, Filiatrault D, Russo P, Lees G, Wilson RD. Outcome of the prenatally diagnosed congenital cystic adenomatoid lung malformation: a Canadian experience. Fetal Diagn Ther. 2001 May-Jun;16(3):178-86. doi: 10.1159/000053905. PMID 11316935
- [Result] Kapralik J, Wayne C, Chan E, Nasr A. Surgical versus conservative management of congenital pulmonary airway malformation in children: A systematic review and meta-analysis. J Pediatr Surg. 2016 Mar;51(3):508-12. doi: 10.1016/j.jpedsurg.2015.11.022. Epub 2015 Dec 9. PMID 26775193
- [Derived] Khan H, Kurup M, Saikia S, Desai A, Mathew M, Sheikh A, Goonasekera CDA. Morbidity after thoracoscopic resection of congenital pulmonary airway malformations (CPAM): single center experience over a decade. Pediatr Surg Int. 2021 May;37(5):549-554. doi: 10.1007/s00383-020-04801-1. Epub 2021 Jan 3. PMID 33388955

DOCUMENTS (1):
  • Informed Consent Form (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04449614/ICF_000.pdf